CLINICAL TRIAL: NCT04380207
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability and Pharmacokinetics of Intravenous (IV) QPX7728 Alone and in Combination With QPX2014 in Healthy Adult Subjects
Brief Title: P1 Single and Multiple Ascending Dose (SAD/MAD) Study of IV QPX7728 Alone and Combined With QPX2014 in NHV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Qpex-200
Record Dates: First submitted 2020-04-21; First posted 2020-05-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Bacterial Infections
Keywords: beta-lactam antibiotic
MeSH Terms: conditions — Bacterial Infections | interventions — QPX7728; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled ascending single, multiple and combination dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, placebo controlled ascending single- and multiple-dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- QPX7728 (Experimental): antibiotic
  Interventions: Drug: QPX7728
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo
- QPX2014 (Experimental): antibiotic
  Interventions: Drug: QPX2014

INTERVENTIONS:
Drug: QPX7728 — antibiotic
  Other Names: IV
  Arms: QPX7728
Drug: Placebo — Placebo comparator
  Other Names: IV saline
  Arms: Placebo
Drug: QPX2014 — antibiotic
  Other Names: IV
  Arms: QPX2014

SUMMARY:
QPX7728 is an ultra-broad-spectrum beta-lactamase inhibitor, with activity against numerous beta-lactamases, including class A extended spectrum beta-lactamases (ESBLs), class C cephalosporinases, and extended spectrum class D oxacillinases (OXA) that can hydrolyze cephalosporins and can be found in Enterobacteriaceae and Pseudomonas aeruginosa (P. aeruginosa). QPX7728 is also a potent inhibitor of carbapenemases from all molecular classes, such as class A Klebsiella pheumoniae carbapenemase (KPC), class B New-Dehli Metalo-beta-lactamase (NDM) and Verona integron-encoded metallo-beta-lactamase (VIM), and class D OXA-48 that are found in carbapenem resistant Enterobacteriaceae, and also class D carbapenemases such as OXA-23 that are found in carbapenem resistant Acinetobacter baumannii.

DETAILED DESCRIPTION:
The Centers for Disease Control (CDC) has listed carbapenem-resistant Enterobacteriaceae and Acinetobacter as urgent threats and multidrug resistant Pseudomonas, and extended spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae as serious threats [CDC, 2019]. Consistent with the global nature of these resistant bacteria, the World Health Organization (WHO) has designated carbapenem-resistant, ESBL-producing Enterobacteriaceae, carbapenem-resistant Acinetobacter baumannii, and carbapenem-resistant Pseudomonas aeruginosa as pathogens for which new agents are critically needed [WHO, 2017].

Qpex Biopharma is developing a fixed combination antibiotic of QPX2014 plus an ultra-broad spectrum beta-lactamase inhibitor, QPX7728.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females of non-child bearing potential, 18 to 55 years of age (inclusive).
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination) as assessed by the PI.
4. Voluntarily consent to participate in the study.
5. If male, agree to be sexually abstinent or agree to use two approved methods of contraception when engaging in sexual activity from study check-in through completion of the end-of-study. Subjects must agree to use two approved methods of contraception for 30 days following the last administration of the study drug, and to not donate sperm during this same period of time. In the event that the sexual partner is surgically sterile, contraception is not necessary.
6. Females of non-childbearing potential with serum follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL are either postmenopausal (defined as 12 months spontaneous amenorrhea) or have undergone sterilization procedures at least 6 months prior to dosing.

Exclusion Criteria:

1. History or presence of significant (based on the PI assessment) cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug/alcohol testing at screening or check-in (Day -1). A repeat test may be performed at the Investigator's discretion in circumstances where a positive result is suspected to be caused by consumption of non-illicit substances.
3. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
4. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
5. Use of more than an average of 5 packs/week of tobacco/nicotine-containing product within 6 months prior to Day 1. Subjects must agree to refrain from smoking for the duration of the study.
6. Excessive intake of alcohol, defined as an average daily intake of greater than 2 standard drinks for women and 4 standard drinks for men, (1 bottle of beer (375mL) is equivalent to approximately 1.4 standard drinks, 1 glass of spirits (30mL) is equivalent to approximately 1 standard drink and 1 glass (150mL) of wine is equivalent to approximately 1.5 standard drinks).
7. Use of any prescription medication (with the exception of hormone replacement therapy for females) within 14 days prior to Day 1.
8. Use of any over-the-counter (OTC) medication, including herbal products, probiotics and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of paracetamol is allowed for acute events at the discretion of the PI.
9. Use of antacids, H2 receptor blockers or proton pump inhibitors 3 days prior to Day 1.
10. Documented hypersensitivity reaction or anaphylaxis to any medication, including beta-lactam antibiotics.
11. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1.
12. Plasma donation within 7 days prior to Day 1.
13. Participation in another investigational clinical trial within 30 days prior to Day 1 or within 5 half-lives of the previous investigational drug, whichever is longer.
14. Surgery within the past three months prior to Day 1 determined by the PI to be clinically relevant.
15. Any significant (based on the PI assessment) acute illness within 30 days prior to Day 1.
16. QTcF interval >450 msec for males and >470 for females or history of prolonged QT syndrome at screening or check-in (Day -1).
17. Calculated creatinine clearance less than 80 mL/min (Cockcroft- Gault method) at screening or check-in (Day -1).
18. Subjects who have any clinically significant abnormalities on laboratory values at screening or check-in (Day -1), in particular:

    1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL.
    2. Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
19. Liver function abnormalities at screening or check-in (Day -1) (defined by an elevation in bilirubin, AST or ALT > ULN of the normal range for subjects based on age and sex).
20. Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment -Emergent Adverse events (AEs) by subject and by cohort (single, multiple and combination dose) | up to 21 days
  Number of patients with Treatment-Emergent AEs by treatment arm, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters (single, multiple and combination dose) | up to 21 days
  Number of patients with changes in safety parameters before and after dosing by subject and treatment arm
Peak plasma Concentration measurements by subject and by cohort (Cmax) (single, multiple and combination dose) | up to 21 days
  Comparison will be performed between the cohorts for Cmax. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Area under the plasma concentration versus time curve (AUC) between cohorts (single, multiple and combination dose) | up to 21 days
  Comparison will be performed between the cohorts for AUC. Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Urine Pharmacokinetic (PK) amount excreted by subject and by cohort (single, multiple and combination dose) | up to 21 days
  Urine PK parameters such as amount excreted will be calculated from urinary excretion data
Urine PK % dose excreted by subject and by cohort (single, multiple and combination dose) | up to 21 days
  Urine PK parameters such as amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (2):
- Altasciences, Cypress, California, United States
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No